CLINICAL TRIAL: NCT05262881
Title: A Retrospective, Observational Study on the Response to Caplacizumab Treatment in aTTP Patients: the Italian Experience (ROSCAPLI)
Acronym: ROSCAPLI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Raimondo De Cristofaro, Professor, Catholic University of the Sacred Heart
Other Study IDs: 4305
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Thrombotic Thrombocytopenic Purpura, Acquired
MeSH Terms: conditions — Thrombotic thrombocytopenic purpura, acquired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter, retrospective, observational study in patients with acquired thrombotic thrombocytopenic purpura (aTTP) treated with plasma exchange (PEX) in association with caplacizumab, and immunosuppression between Q4-2019 and 28 February2021. The retrospective study will measure: Age, sex, BMI, blood pressure at diagnosis, Platelet count at diagnosis and at the follow up visits, Hb level at diagnosis at the follow up visits, White blood cell count at diagnosis at the follow up visits, Creatinine at diagnosis at the follow up visits, schistocytes count at diagnosis at the follow up visits, LDH at diagnosis at the follow up visits, Coombs' assay at diagnosis, alanine-leucine-amino-transferase (ALT) at diagnosis at the follow up visits, total bilirubin at diagnosis at the follow up visits, Troponin above ULN at any point, ADAMTS13 activity (where measured) at diagnosis at the follow up visits, Anti-ADAMTS13 antibodies (where measured) at diagnosis at the follow up visits.

The primary objective in this study is the description and quantification of clinical response in terms of platelet count recovery in patients with aTTP treated t with caplacizumab , in addition to PEX and immunosuppression in the real-world setting. The secondary objectives include: number of exacerbations, defined as recurrent thrombocytopenia within 30 days after the end of therapy; rate of relapse, defined as a TTP event occurring more than 30 days after the end of daily plasma exchange; refractoriness; defined by the lack of a doubling of platelet count after 4 days of treatment and a lactate dehydrogenase level that remained above the upper limit of the normal range, TTP-related mortality and evaluation of adverse events.

DETAILED DESCRIPTION:
This study is a multicenter, retrospective, observational study in patients with acquired thrombotic thrombocytopenic purpura (aTTP) treated with plasma exchange (PEX) in association with caplacizumab, and immunosuppression between Q4-2019 and 28 February2021.

Study design

The retrospective study will measure the following vital, clinical chemistry, hematological, and hemostatic parameters, according to the consensus guidelines of aTTP diagnosis and as a part of routine diagnostic work-up:

* Age, sex, BMI, blood pressure at diagnosis
* Platelet count at diagnosis and at the follow up visits
* Hb level at diagnosis at the follow up visits
* White blood cell count at diagnosis at the follow up visits
* Creatinine at diagnosis at the follow up visits
* schistocytes count at diagnosis at the follow up visits
* LDH at diagnosis at the follow up visits
* Coombs' assay at diagnosis
* alanine-leucine-amino-transferase (ALT) at diagnosis at the follow up visits
* total bilirubin at diagnosis at the follow up visits
* Troponin above ULN at any point
* ADAMTS13 activity (where measured) at diagnosis at the follow up visits
* Anti-ADAMTS13 antibodies (where measured) at diagnosis at the follow up visits The clinical signs will be parametrized by the PLASMIC score and the Glasgow score, where calculated in the various centers. The PLASMIC score and the Glasgow score will be evaluated according to the obtained values (0-4, 5-6, and 7; <13 and 13-15, respectively). All the clinical and laboratory parameters will be taken in each center and reported in the CRF.

OBJECTIVES The primary objective in this study is the description and quantification of clinical response in terms of platelet count recovery in patients with aTTP treated t with caplacizumab , in addition to PEX and immunosuppression in the real-world setting. The Secondary objectives include: Number of exacerbations, defined as recurrent thrombocytopenia within 30 days after the end of therapy; Rate of relapse, defined as a TTP event occurring more than 30 days after the end of daily plasma exchange;Refractoriness; defined by the lack of a doubling of platelet count after 4 days of treatment and a lactate dehydrogenase level that remained above the upper limit of the normal range, TTP-related mortality and evaluation of adverse events.

Data collection and management A customized eCRF (RedCap) will be created for the study and only the principal investigator and collaborating investigators of the center will have access to patient medical records during the study.

STATISTICAL CONSIDERATIONS Qualitative variables will be expressed by absolute and percentage frequency. Quantitative variables will be previously assessed for their distribution by the Shapiro-Wilk test. Normally distributed data will be described by mean and standard deviation (SD), whilst non-normally distributed variable by median and interquartile range (IQR).

INFORMED CONSENT Informed consent form will be collected for all except for all patients whom death is ascertained

ELIGIBILITY:
Inclusion Criteria:

* The patients included in this study should have received caplacizumab for treatment in the period between Q4-2019 and the end of February 2021 while the end of follow up observation is scheduled for Q1-2021 (to observe at least one month of post treatment follow up). The diagnosis should be based on either clinical/laboratory parameters inclusive of measurement of ADAMTS13 level <10%) or the PLASMIC score (platelets, lysis, active cancer, stem cell or solid organ transplant, MCV, INR, and creatinine) with intermediate and high risk (sore>5) already computed or retrospectively calculated as previously detailed for centers that did not measure the ADAMTS13 level.

Exclusion Criteria:

* Patients treated with uncertain aTTP diagnosis according to the above inclusion criteria and manifesting clinical signs like aTTP but characterized by a different pathogenesis (e.g. cancer, sepsis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients treated for acute aTTP episodes in the hematology, internal medicine, and critical care centers between Q4-2019 and Q1-2021 in Italy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Time-to-response of Treatment Defined by a Confirmed Recovery of Platelets | 18 months
  Platelet response was defined as recovery of platelets ≥ 150,000/µL.

SECONDARY OUTCOMES:
study of critical parameters | 18 months
  1. Number and percentage of subjects with TTP-Related Death
  2. Number and percentage of subjects with relapse of TTP, defined as a TTP event occurring more than 30 days after the end of daily plasma exchanges
  3. assessment of all SAEs of thromboembolic events
  4. Number and percentage of subjects with exacerbations, defined as recurrent thrombocytopenia within 30 days after the end of daily plasma exchanges that required reinitiation of daily exchanges
  5. Number and percentage of subjects with refractory TTP (); and the time to normalization (i.e., to a level below the defined upper limit of the normal range) of three organ-damage markers (LDH, cardiac troponin I, and serum creatinine).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Scully M, Hunt BJ, Benjamin S, Liesner R, Rose P, Peyvandi F, Cheung B, Machin SJ; British Committee for Standards in Haematology. Guidelines on the diagnosis and management of thrombotic thrombocytopenic purpura and other thrombotic microangiopathies. Br J Haematol. 2012 Aug;158(3):323-35. doi: 10.1111/j.1365-2141.2012.09167.x. Epub 2012 May 25. No abstract available. PMID 22624596
- [Result] Rizzo C, Rizzo S, Scire E, Di Bona D, Ingrassia C, Franco G, Bono R, Quintini G, Caruso C. Thrombotic thrombocytopenic purpura: a review of the literature in the light of our experience with plasma exchange. Blood Transfus. 2012 Oct;10(4):521-32. doi: 10.2450/2012.0122-11. Epub 2012 Jun 27. No abstract available. PMID 22790258
- [Result] Bell WR, Braine HG, Ness PM, Kickler TS. Improved survival in thrombotic thrombocytopenic purpura-hemolytic uremic syndrome. Clinical experience in 108 patients. N Engl J Med. 1991 Aug 8;325(6):398-403. doi: 10.1056/NEJM199108083250605. PMID 2062331
- [Result] Nguyen L, Li X, Duvall D, Terrell DR, Vesely SK, George JN. Twice-daily plasma exchange for patients with refractory thrombotic thrombocytopenic purpura: the experience of the Oklahoma Registry, 1989 through 2006. Transfusion. 2008 Feb;48(2):349-57. doi: 10.1111/j.1537-2995.2007.01530.x. Epub 2007 Nov 19. PMID 18028271
- [Result] Balduini CL, Gugliotta L, Luppi M, Laurenti L, Klersy C, Pieresca C, Quintini G, Iuliano F, Re R, Spedini P, Vianelli N, Zaccaria A, Pogliani EM, Musso R, Bobbio Pallavicini E, Quarta G, Galieni P, Fragasso A, Casella G, Noris P, Ascari E; Italian TTP Study Group. High versus standard dose methylprednisolone in the acute phase of idiopathic thrombotic thrombocytopenic purpura: a randomized study. Ann Hematol. 2010 Jun;89(6):591-6. doi: 10.1007/s00277-009-0877-5. Epub 2009 Dec 23. PMID 20033409
- [Result] Ziman A, Mitri M, Klapper E, Pepkowitz SH, Goldfinger D. Combination vincristine and plasma exchange as initial therapy in patients with thrombotic thrombocytopenic purpura: one institution's experience and review of the literature. Transfusion. 2005 Jan;45(1):41-9. doi: 10.1111/j.1537-2995.2005.03146.x. PMID 15647017
- [Result] Beloncle F, Buffet M, Coindre JP, Munoz-Bongrand N, Malot S, Pene F, Mira JP, Galicier L, Guidet B, Baudel JL, Subra JF, Tanguy-Schmidt A, Pourrat J, Azoulay E, Veyradier A, Coppo P; Thrombotic Microangiopathies Reference Center. Splenectomy and/or cyclophosphamide as salvage therapies in thrombotic thrombocytopenic purpura: the French TMA Reference Center experience. Transfusion. 2012 Nov;52(11):2436-44. doi: 10.1111/j.1537-2995.2012.03578.x. Epub 2012 Mar 8. PMID 22404639
- [Result] Sayani FA, Abrams CS. How I treat refractory thrombotic thrombocytopenic purpura. Blood. 2015 Jun 18;125(25):3860-7. doi: 10.1182/blood-2014-11-551580. Epub 2015 Mar 17. PMID 25784681
- [Result] Lim W, Vesely SK, George JN. The role of rituximab in the management of patients with acquired thrombotic thrombocytopenic purpura. Blood. 2015 Mar 5;125(10):1526-31. doi: 10.1182/blood-2014-10-559211. Epub 2015 Jan 8. No abstract available. PMID 25573992
- [Result] Vazquez-Mellado A, Pequeno-Luevano M, Cantu-Rodriguez OG, Villarreal-Martinez L, Jaime-Perez JC, Gomez-De-Leon A, De La Garza-Salazar F, Gonzalez-Llano O, Colunga-Pedraza P, Sotomayor-Duque G, Gomez-Almaguer D. More about low-dose rituximab and plasma exchange as front-line therapy for patients with thrombotic thrombocytopenic purpura. Hematology. 2016 Jun;21(5):311-6. doi: 10.1080/10245332.2015.1133008. Epub 2016 Feb 24. PMID 26907228
- [Result] Scully M, McDonald V, Cavenagh J, Hunt BJ, Longair I, Cohen H, Machin SJ. A phase 2 study of the safety and efficacy of rituximab with plasma exchange in acute acquired thrombotic thrombocytopenic purpura. Blood. 2011 Aug 18;118(7):1746-53. doi: 10.1182/blood-2011-03-341131. Epub 2011 Jun 2. PMID 21636861
- [Result] Page EE, Kremer Hovinga JA, Terrell DR, Vesely SK, George JN. Rituximab reduces risk for relapse in patients with thrombotic thrombocytopenic purpura. Blood. 2016 Jun 16;127(24):3092-4. doi: 10.1182/blood-2016-03-703827. Epub 2016 Apr 8. No abstract available. PMID 27060171
- [Result] Hie M, Gay J, Galicier L, Provot F, Presne C, Poullin P, Bonmarchand G, Wynckel A, Benhamou Y, Vanhille P, Servais A, Bordessoule D, Coindre JP, Hamidou M, Vernant JP, Veyradier A, Coppo P; French Thrombotic Microangiopathies Reference Centre. Preemptive rituximab infusions after remission efficiently prevent relapses in acquired thrombotic thrombocytopenic purpura. Blood. 2014 Jul 10;124(2):204-10. doi: 10.1182/blood-2014-01-550244. Epub 2014 May 28. PMID 24869941
- [Result] Rottenstreich A, Hochberg-Klein S, Rund D, Kalish Y. The role of N-acetylcysteine in the treatment of thrombotic thrombocytopenic purpura. J Thromb Thrombolysis. 2016 May;41(4):678-83. doi: 10.1007/s11239-015-1259-6. PMID 26245827
- [Result] Eskazan AE. Bortezomib therapy in patients with relapsed/refractory acquired thrombotic thrombocytopenic purpura. Ann Hematol. 2016 Oct;95(11):1751-6. doi: 10.1007/s00277-016-2804-x. Epub 2016 Sep 3. PMID 27590601
- [Result] Masias C, Cataland SR. Novel therapies in thrombotic thrombocytopenic purpura. Res Pract Thromb Haemost. 2017 Dec 18;2(1):19-26. doi: 10.1002/rth2.12066. eCollection 2018 Jan. PMID 30046703
- [Result] Volker LA, Kaufeld J, Miesbach W, Brahler S, Reinhardt M, Kuhne L, Muhlfeld A, Schreiber A, Gaedeke J, Tolle M, Jabs WJ, Ozcan F, Markau S, Girndt M, Bauer F, Westhoff TH, Felten H, Hausberg M, Brand M, Gerth J, Bieringer M, Bommer M, Zschiedrich S, Schneider J, Elitok S, Gawlik A, Gackler A, Kribben A, Schwenger V, Schoenermarck U, Roeder M, Radermacher J, Bramstedt J, Morgner A, Herbst R, Harth A, Potthoff SA, von Auer C, Wendt R, Christ H, Brinkkoetter PT, Menne J. Real-world data confirm the effectiveness of caplacizumab in acquired thrombotic thrombocytopenic purpura. Blood Adv. 2020 Jul 14;4(13):3085-3092. doi: 10.1182/bloodadvances.2020001973. PMID 32634236
- [Result] Jamme M, Rondeau E. The PLASMIC score for thrombotic thrombocytopenic purpura. Lancet Haematol. 2017 Apr;4(4):e148-e149. doi: 10.1016/S2352-3026(17)30024-8. Epub 2017 Mar 2. No abstract available. PMID 28259521
- See also: European-Medicines-Agency. Cablivi (caplacizumab): summary of product characteristics. Document of the European Medicines Agency. 2018; — http://www.ema.europa.eu.